CLINICAL TRIAL: NCT04304677
Title: Development of Automated Algorithm Detecting Physiologic Major Stenosis and Its Relationship With Post-PCI Clinical Outcomes (Algorithm-PCI)
Brief Title: Automated Algorithm Detecting Physiologic Major Stenosis and Its Relationship With Post-PCI Clinical Outcomes
Acronym: Algorithm-PCI
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: Inje University Ilsan Paik Hospital (Other); Keimyung University Dongsan Medical Center (Other); Ulsan University Hospital (Other); Sejong General Hospital (Other); Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Joo Myung Lee, Assistant Professor, Samsung Medical Center
Other Study IDs: Algorithm20200211
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Ischemic Heart Disease
Keywords: fractional flow reserve; delta FFR per unit time; percutaneous coronary intervention; prognosis
MeSH Terms: conditions — Myocardial Ischemia | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pre PCI state: The current study will analyze the pre-PCI pullback recording and amount of FFR step-up. The association of the amount of FFR step-up with post-PCI percent FFR increase, post-PCI FFR, and clinical outcome at 2 years will be analyzed
  Interventions: Device: Percutaneous coronary intervention

INTERVENTIONS:
Device: Percutaneous coronary intervention — 1. Pre-PCI FFR pullback recording was done with conventional system
  2. Automated algorithm to calculate delta FFR per unit time was developed
  3. PCI was performed using 2nd generation DES
  Other Names: Fractional flow reserve

SUMMARY:
The presence of myocardial ischemia is the most important prognostic indicator in patients with coronary artery disease. Therefore, the purpose of percutaneous coronary intervention (PCI) is to relieve myocardial ischemia caused by the target stenosis. Fractional flow reserve (FFR) is an invasive physiologic index used to define functionally significant coronary stenosis, and its prognostic implications are supported by numerous studies. Contrary to the clear cutoff value and the benefit of FFR in pre-PCI evaluation, there have been various results regarding optimal cut-off values for post-PCI FFR. Nevertheless, the positive association between post-PCI FFR and the risk of future events has been reproduced by several studies.

PCI with stent implantation is basically a local treatment and post-PCI FFR reflects both residual stenosis in the stented segment and remaining disease beyond the stented segment in the target vessel(s).

Therefore, post-PCI FFR alone cannot fully discriminate the degree of contribution of each component. The relative increase of FFR with PCI is determined by the interaction of baseline severity of a target lesion, baseline disease burden of a target vessel, adequacy of PCI and residual disease burden in a target vessel.

However, the most important problem in stratifying patients with better expected post-PCI physiologic results and following clinical outcome would be that there has been no clear method to identify these patients in pre-PCI phase.

In this regard, we hypothesized that the amount of FFR step-up in pre-PCI pullback recording would determine the physiologic nature of target stenosis. For example, stenosis with sufficient step-up of FFR would deserve local treatment with PCI and these lesions would result in higher percent FFR increase, post-PCI FFR, and better clinical outcome than those without sufficient amount of FFR step-up.

For this, we sought to develop automated algorithm to define physiologic major stenosis versus minor stenosis using pre-PCI pullback recording.

DETAILED DESCRIPTION:
The current study cohort consisted with 3 cohort. In order to derive and validate the optimal cut-off values of FFR step-up amount for physiologic major vs minor stenosis and for physiologic minor stenosis vs. signal noise, the below 3 cohorts will be used.

1. Derivation cohort of defining the optimal cut off value of FFR step-up amount for physiologic major vs minor stenosis and for physiologic minor stenosis vs. signal noise.

   The cohort of no coronary atherosclerosis confirmed by both angiography and intravascular ultrasound will be derived from patients with heart transplantation (NCT02798731).

   The cohort of significant focal or diffuse obstructive coronary artery disease with functional significance defined by FFR<=0.80 will be derived from post-PCI registry of Samsung Medical Center.
2. Internal validation cohort will be post-PCI registry of Samsung Medical Center which enrolled 236 patients who underwent both pre- and post-PCI physiologic assessment after angiographically successful PCI using 2nd generation drug-eluting stent. Among this cohort, 234 patients with available pre-PCI pullback recording will be analyzed.
3. External validation cohort will be COE-PERSPECTIVE registry (NCT01873560) which enrolled patients who underwent PCI for lesions with FFR<=0.80 and underwent post-PCI physiologic assessment.

Among the 835 patients, 252 patients with available pre-PCI pullback recording will be analyzed.

For the association between physiologic major, minor, or mixed stenosis classified using the optimal cut-off values of FFR step-up amount for physiologic major vs minor stenosis and for physiologic minor stenosis vs. signal noise, the patient level pooled data of both Samsung Medical Center registry and COE-PERSPECTIVE registry will be used.

ELIGIBILITY:
Inclusion Criteria:

* any patient meets eligible criteria who underwent PCI with DES followed by invasive physiologic assessment at the index procedure
* any patient who underwent PCI for lesions with pre-PCI FFR<=0.80
* available pre-PCI FFR pullback recording
* available both post-PCI FFR measurement

Exclusion Criteria:

* unavailable pre-PCI FFR pullback recording
* unavailable post-PCI FFR measurement
* culprit vessel of acute coronary syndrome
* failed achieving TIMI 3 flow at the end of PCI
* left ventricular ejection fraction <30%
* graft vessel
* collateral feeder
* in-stent restenosis
* primary myocardial or valvular heart disease
* in patient whose life expectancy less than 2 years
* visible thrombus of target vessel segment

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who diagnosed obstructive coronary artery disease and evaluated by pre-PCI FFR measurement and pullback recording, then treated by DES with invasive physiologic evaluation at the index procedure.
Sampling Method: Non-Probability Sample
Enrollment: 486 (Estimated)
Dates: Start 2016-03-22 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Percent FFR increase after PCI | Immediate post-PCI
  ([Post-PCI FFR - Pre-PCI FFR]/Pre-PCI FFR * 100)
Post-PCI FFR | Immediate post-PCI
  FFR value measured after angiographically successful PCI

SECONDARY OUTCOMES:
Target Vessel Failure | 2 years after index procedure
  a composite of cardiac death, clinically-driven target vessel-related myocardial infarction, and clinically-driven target vessel revascularization. The target vessel will be defined as the treated vessel with 2nd generation DES which was assessed by post stent fractional flow reserve.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
De-identified patient data will be shared upon reasonable request after discussion in executive committee and developer of algorithm.

REFERENCES:
- [Derived] Shin D, Dai N, Lee SH, Choi KH, Lefieux A, Molony D, Hwang D, Kim HK, Jeon KH, Lee HJ, Jang HJ, Ha SJ, Park TK, Yang JH, Song YB, Hahn JY, Choi SH, Doh JH, Shin ES, Nam CW, Koo BK, Gwon HC, Ge J, Lee JM. Physiological Distribution and Local Severity of Coronary Artery Disease and Outcomes After Percutaneous Coronary Intervention. JACC Cardiovasc Interv. 2021 Aug 23;14(16):1771-1785. doi: 10.1016/j.jcin.2021.06.013. PMID 34412795
- [Derived] Lee SH, Shin D, Lee JM, Lefieux A, Molony D, Choi KH, Hwang D, Lee HJ, Jang HJ, Kim HK, Ha SJ, Kwak JJ, Park TK, Yang JH, Song YB, Hahn JY, Doh JH, Shin ES, Nam CW, Koo BK, Choi SH, Gwon HC. Automated Algorithm Using Pre-Intervention Fractional Flow Reserve Pullback Curve to Predict Post-Intervention Physiological Results. JACC Cardiovasc Interv. 2020 Nov 23;13(22):2670-2684. doi: 10.1016/j.jcin.2020.06.062. Epub 2020 Oct 14. PMID 33069650